CLINICAL TRIAL: NCT06116331
Title: The Mind-Body IBD Study: Understanding the Bidirectional Relationship Between Depression and Anxiety With Physical Health Outcomes and Inflammation
Brief Title: The Mind-Body IBD Study: Understanding the Mind-body Connection in IBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: 33844
Record Dates: First submitted 2023-10-25; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Crohn Colitis
Keywords: mental health; depression; anxiety; psychology; health; exercise; stress; diet; sleep; adherence
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Psychological Well-Being; Depression; Anxiety Disorders; Motor Activity | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants will complete 3 online questionnaires at 6 month intervals. At the first two time points they will also be asked to submit 2 at home stool sample tests, to assess fecal calprotectin.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Participants will answer questionnaires and submit stool samples.

SUMMARY:
An aspect of IBD care that is often overlooked is mental health treatment. Common mental health problems, such as anxiety and depression are very common in IBD, with a meta-analysis estimating prevalence as high as 25.2% for depression and 32.1% for anxiety. The prevalence of anxiety and depression increases when individuals with active disease are considered, with rates as high as 57.6% for anxiety and 38.9% for depression. Comorbid depression and anxiety in IBD is associated with greater symptom severity, even when statistically controlling for disease activity; more frequent and expensive emergency department visits and inpatient stays, higher costs relating to IBD-related surgery, medication and personal expenditure; noncompliance with medical treatment and finally, increased likelihood of experiencing flares.

However, very few studies attempt to unpick the precise mechanism of these bidirectional relationships.

Indeed, depression and anxiety may have direct effects on physical health through inflammatory or psychoneuroimmunological pathways. Very few studies investigate the longitudinal brain-gut relationship with regards to objective measures of inflammation. Additionally, the indirect effects of mental health are often overlooked. Depression and anxiety are routinely associated with health behaviours, such as diet, physical activity, sleep, and tobacco/alcohol use.These health behaviours are important factors, given their impact on physical health outcomes. Therefore, a thorough investigation is required to ascertain the precise mechanisms that underpin the bidirectional relationship between depression/anxiety and inflammation/physical health, as this will enable practitioners and researchers to establish non-invasive, behavioural treatment targets for this patient group.

AIM The broad aim of this project is to explore whether anxiety/depression has a direct or indirect (via health behaviours) on i) inflammation levels ii) clinical activity and iii) healthcare usage at follow-up, in a population of IBD patients. A secondary aim of the project will be to explore whether changes in disease activity, as measured by self-report measures and faecal calprotectin, explains changes in anxiety and depression symptoms at follow up.

DETAILED DESCRIPTION:
Participants will be asked to answer online questionnaires at 3 time points, 6 months apart. They will also be asked to do an at-home stool sample test at the first two time points.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported diagnosis of IBD (pseudo-confirmed with participant's self-reported IBD medication or medication history)
2. Willing and able to give informed consent and participate in the study
3. Aged 18 and over
4. Sufficient command of written and spoken English to understand study procedures and documents, and complete self-report questionnaires
5. UK resident (GP registered)
6. Email address, telephone number and postal address to enable all study procedures
7. Experience at least one flare (requiring medical escalation or medication change) within the last two years

Exclusion Criteria:

1. Under 18 years
2. Lives outside of the UK
3. Insufficient command of English to understand study documents and procedures
4. Not able to give informed consent Regular use of non-steroidal anti-inflammatory drugs (NSAIDs) in the last two weeks.
5. People with a cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with IBD in the UK, who have experienced a flare within the last 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychological distress: Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Month 0, Month 6, Month 12
  The PHQ-ADS is a composite measure of the Generalised Anxiety Disorder questionnaire (GAD-7) and the Patient Health Questionnaire (PHQ-9). Min score = 0, Max score = 48, with higher scores indicating higher levels of distress.
Depression: Patient Health Questionnaire - (PHQ-9) | Month 0, Month 6, Month 12
  Depression. Min score = 0, Max score = 27, with higher scores indicating greater depression.
Anxiety: Generalised Anxiety Disorder scale (GAD-7) | Month 0, Month 6, Month 12
  Anxiety. Min score = 0, Max score = 21, with higher scores indicating greater anxiety
Fecal Calprotectin | Month 0, Month 6
  Measure of intestinal inflammation, higher levels indicate greater inflammation.
Health service use | Month 0, Month 6, Month 12
  4 service use items (GP, psychologist, emergency care, secondary care service) from the client service receipt inventory (CSRI) will be used. Frequency and duration of particular services will be recorded, from which a total time will be calculated. There is no maximum value. Higher scores indicate more health service time used.
IBD activity | Month 0, Month 6, Month 12
  For Crohn's Disease patients: The Patient-Reported Outcomes for the Assessment of Crohn's Disease Activity (PRO-CD). The scale contains two sub-scales: 1) bowel signs and symptoms, 2) functional symptoms. Each scale is scored separately. There is no total score for the PRO-CD. The first sub-scale starts at 0 and has no maximum value, with greater scores indicating greater bowel signs/symptoms. The second subscale ranges from 0-21, with higher scores indicating greater functional symptoms.
  For Ulcerative Colitis / unclassified patients: The Patient-Reported Outcomes for Assessment of Ulcerative Colitis (PRO-UC). The scale has 9-items and includes two scales: 1) Bowel signs/symptoms and 2) functional symptoms. The first sub-scale starts at 0 and has no maximum value, with greater scores indicating greater bowel signs/symptoms. The second subscale ranges from 0-21, with higher scores indicating greater functional symptoms.

SECONDARY OUTCOMES:
Body Mass Index | Month 0, Month 6, Month 12
  Weight (in kg) and Height (in m) will be combined to calculate BMI (weight in kg / (height in m)^2
Smoking status | Month 0, Month 6, Month 12
  Current smoking status, including amount of cigarettes consumed per day.
Alcohol Consumption | Month 0, Month 6, Month 12
  Number of units drunk in the past week.
Physical activity: International Physical Activity Questionnaire | Month 0, Month 6, Month 12
  Physical activity. There are three subscales (vigorous activity, moderate activity and lower-level activity). Scores will be in minutes. Higher scores will indicate more physical activity performed.
IBD medication | Month 0, Month 6, Month 12
  Current medication and dose.
IBD flares | Month 0, Month 6, Month 12
  Frequency and severity (4-point scale) of IBD flares (in last 6 months)
Sleep - the Pittsburgh Sleep Quality Index (PSQI) | Month 0, Month 6, Month 12
  Sleep quality in the last month. Min=0, max=21, with higher scores indicating worse sleep quality.
Diet - Healthy Eating Assessment | Month 0, Month 6, Month 12
  8-item simplified food frequency questionnaire designed for use in primary care settings. The tool will be adapted so that each item is score 1-5. Mix=8, max=40, with higher scores indicating better diet quality.
IBD quality of life - short Inflammatory Bowel Disease Questionnaire (sIBDQ) | Month 0, Month 6, Month 12
  The sIBDQ is a ten-item questionnaire that covers four domains: bowel symptoms, systemic symptoms, emotional health, and social functions. Min=10, max=70, with a lower score indicating lower quality of life.
Medication Adherence - Medication Adherence Report Scale (MARS) | Month 0, Month 6, Month 12
  5-item scale on a 5-point scale.Mix=0, Max=20, with higher scores indicating better adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Rona Moss-Morris, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study information and sign up — https://linktr.ee/mindbodyibdstudy